CLINICAL TRIAL: NCT06475794
Title: Investigation of Q Angle and Related Factors in Osteoporosis Patients
Brief Title: Investigation of Q Angle in Osteoporosis Patients
Status: Recruiting | Type: Observational
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Head of Physiotherapy and Rehabilitation Department, Firat University
Other Study IDs: 2024/07-33
Record Dates: First submitted 2024-06-14; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Osteopenia; Q angle
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with osteoporosis group: Osteoporosis patients will be evaluated in terms of pain, foot posture, Q angle and lower limbs muscle strength.
  Interventions: Other: Patients with osteoporosis group
- Patients with osteoarthritis group: Osteoarthritis patients will be evaluated in terms of pain, foot posture, Q angle and lower limbs muscle strength.
  Interventions: Other: Patients with osteoarthritis group

INTERVENTIONS:
Other: Patients with osteoporosis group — Pain, Q angle, muscle strength and foot posture will be evaluated.
  Groups: Patients with osteoporosis group
Other: Patients with osteoarthritis group — Osteoarthritis patients will be evaluated in terms of pain, foot posture, Q angle and lower limbs muscle strength.
  Groups: Patients with osteoarthritis group

SUMMARY:
Osteoporosis (OP) is a bone disease characterized by reduced bone density and deterioration of bone tissue, leading to an increased risk of fractures. There are no studies evaluating Q angle in patients with OP and Osteopenia (OPN) in the literature. Therefore, the aim of this study was to examine the Q angle in patients diagnosed with OP and OPN and to compare it with patients diagnosed with OA. The study will be carried out by measuring the Q angle measurement with a goniometer. Pain assessment will be done with Visual Analog Scale (VAS). Lower extremity muscle strength will be assessed with the Medical Research Council (MRC) Scale. Foot posture will be assessed with the Foot Posture Index (FPI).

DETAILED DESCRIPTION:
Osteoporosis (OP) is a bone disease characterized by reduced bone density and deterioration of bone tissue, leading to an increased risk of fractures. According to Calis et al; it was found that patients with hip fracture had a significantly higher Q angle compared to patients without hip fracture. According to You et al; contraction of the quadriceps muscles corrects the Q angle, therefore sports that use high amounts of quadriceps (strength) training are associated with lower Q angles due to the pulling effect of the quadriceps muscle. There are no studies evaluating Q angle in patients with OP and Osteopenia (OPN) in the literature. Therefore, the aim of this study was to examine the Q angle in patients diagnosed with OP and OPN and to compare it with patients diagnosed with OA. The study will be carried out by measuring the Q angle measurement with a goniometer. Pain assessment will be done with Visual Analog Scale (VAS). Lower extremity muscle strength will be assessed with the Medical Research Council (MRC) Scale. Foot posture will be assessed with the Foot Posture Index (FPI).

ELIGIBILITY:
Inclusion Criteria:

* Be willing to participate in the study.
* Being between the ages of 40-65.
* Being a woman.

Exclusion Criteria:

* Patellofemoral abnormalities during examination.
* Acute traumatic patellofemoral dislocations
* Surgical revision around the knee
* History of any previous lower extremity surgery
* Serious trauma

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are willing to participate in the study, being between the ages of 40-65 will be included in the study. Patients who have patellofemoral abnormalities during examination, acute traumatic patellofemoral dislocations, surgical revision around the knee, history of any previous lower extremity surgery and serious trauma will be excluded from the study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Q angle assessment | 1 minute
  Q angle will be evaluated with goniometer.

SECONDARY OUTCOMES:
Pain assessment | 1 minute
  Pain assessment will be done with the Visual Analog Scale (VAS). This measurement is performed with a chart in which no pain is written on one end and very severe pain is written on the other end.
Muscle strength assessment | 2 minutes
  Lower extremity muscle strength will be assessed with the Medical Research Council (MRC) Scale. Muscle strength is graded on a scale of 0 to 5 according to muscle tone and ability to resist the force of gravity.
Foot posture assessment | 1 minute
  Foot posture will be evaluated with the Foot Posture Index (FPI). API is an easy-to-apply, valid and reliable method that provides information about the degree of pronation and supination of the foot with a single numerical result and evaluates the foot in a multidimensional and comprehensive manner.

CONTACTS AND LOCATIONS:
Locations (1):
- Songul Baglan Yentur, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No